CLINICAL TRIAL: NCT01503411
Title: High Resolution Optical Imaging of Barrett's Esophagus Using Nvision Volumetric Laser Endomicroscopy (VLE)
Status: Completed | Type: Observational
Sponsor: NinePoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol No. 11_01
Record Dates: First submitted 2011-12-27; First posted 2012-01-04 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this clinical trial is to evaluate the performance of the Nvision Volumetric Laser Endomicroscopy (VLE) system to visualize subsurface tissue in subjects undergoing esophagogastroduodenoscopy (EGD) and to identify work-flow and training implications for introducing this new imaging modality.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years.
* Patients with either suspected BE presenting for endoscopy or patients with documented BE presenting for follow-up endoscopy likely to require a biopsy or patients presenting for endoscopy for non-BE related conditions other than esophageal varices.
* Ability to provide written, informed consent.
* Females who are able to become pregnant, are willing to take a pregnancy test.

Exclusion Criteria:

* Patients on anticoagulation undergoing high risk procedures in accordance to American Society For Gastrointestinal Endoscopy (ASGE) guideline for the management of antithrombotic agents for endoscopic procedures (2009).
* Patients with esophageal varices that preclude biopsies.
* Presence of an esophageal mass that precludes full distention of the balloon from the Nvision balloon guide sheath.
* Patients with esophageal strictures that would prevent adequate expansion of the balloon from the Nvision balloon guide sheath.
* Patients with known inflammatory disease, esophageal tears or ulcers, which would prohibit full distention of the balloon from the Nvision balloon guide sheath.
* Patients with known eosinophilic esophagitis.
* Patients that are pregnant.
* Patients with a history of hemostasis disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females >18 years of age undergoing esophagogastroduodenoscopy (EGD) for suspected or confirmed Barrett's esophagus (BE)or for non-BE related conditions other than esophageal varices.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | The research participants will be followed and evaluated for the duration of their VLE procedure, an expected average of 10 additional minutes beyond the standard EDG procedure.
  The primary endpoint will be the number of subjects achieving completed VLE imaging studies at the time of EDG.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert C. Wolfsen, MD, Study Chair — Mayo Clinic; Prateek Sharma, MD, Principal Investigator — University Medical Center, Kansas City, MO; Kenneth Wang, MD, Principal Investigator — Mayo Clinic, Rochester, MN; Herbert C Wolfsen, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Massachusetts
  - VA Medical Center, Kansas City, Missouri